CLINICAL TRIAL: NCT03804099
Title: The Effect of Intravitreal Aflibercept on Ocular Perfusion - a Pilot Study
Brief Title: Effect Aflibercept on Ocular Perfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-05.01
Record Dates: First submitted 2018-06-29; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Macular Degeneration; Anti Vascular Endothelial Growth Factor
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — After instillation of topical anesthetic, sterilization of the eyelid, and instillation of 1.25% povidone-iodine drops, 2.0 mg/0.05 mL of aflibercept (Eylea) is injected into the vitreous cavity through a standard pars plana approach (3.5 mm posterior to the limbus) under sterile conditions

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible visual impairment in Western Countries. It is a well-established fact that vascular endothelial growth factor (VEGF) plays a key part in the development of the neovascular (or exsudative) form of AMD. Today, VEGF-inhibition by means of injection of anti-VEGF agents into the vitreous cavity constitutes the gold standard of AMD therapy. In physiological conditions, VEGF acts as a vasodilator by activating endothelial nitric oxide synthase. As a consequence, VEGF inhibition should result in significant ocular vasoconstriction, which has in fact been demonstrated for bevacizumab and ranibizumab, two of the three available VEGF-inhibitors. The understanding and awareness of potentially harmful implications of the induced vasoconstriction on retinal and/or optic nerve head structure and function is sparse. This is especially delicate, as most patients with exsudative AMD require repeated injections on a monthly basis for many years. Aflibercept, the latest anti-VEGF agent approved for intravitreal use in 2011, offers a superior binding affinity for VEGF compared to the former two drugs. However, as of today, its effect on ocular circulation is unclear. With Laser Speckle Flowgraphy (LSFG), a commercially available, non-invasive and patient-friendly method for the evaluation of blood flow at the optic nerve head, the choroid and retina has arisen in recent years.

We aim to measure ocular perfusion with LSFG before and after 3 consecutive injections of aflibercept in unilateral neovascular age-related maculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 50 years
* written informed consent for participation in the study
* Scheduled for 3 consecutive intravitreal injections (4 week intervals) of aflibercept for treatment of exudative AMD in one eye
* Subject is generally healthy with no current significant or a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination. A significant disorder is defined as a disease or medical condition associated with impaired health status, requiring regular or current medical treatment and/or follow up. For the purposes of this study, an investigator may classify a medical condition as a nonsignificant disorder despite the fact that the subject receives treatment. Subjects having controlled Stage 1 hypertension (blood pressure of 140-159 mmHg systolic and/or 90-99 mmHg diastolic) are eligible for participation in this study.
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Active exudative AMD requiring treatment of both eyes
* Ocular surgery (including intravitreal injection) during the 3 months preceding the study
* Vitrectomized eyes
* Ametropia > 6 Dpt
* Relevant ophthalmic diseases/conditions that could interfere with LSFG measurements (e.g. glaucoma, optic nerve head drusen, tilted disc, etc.)
* Ocular infection or clinically significant inflammation
* Opacities of the cornea (e.g. corneal scars, corneal oedema), the lens (e.g. LOCS-II grading > 2, posterior capsule opacification) or the vitreous (e.g. vitreous haemorrhage, asteroid hyalosis)
* Patients who are not able to cooperate or with insufficient ability to fixate (tremor, nystagmus)
* Blood donation in the 3 weeks preceding the study
* Participation in a clinical trial in the 3 weeks preceding the study
* Pre- or perimenopausal women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Mean blur ratio (LSFG) | Baseline, 1 week (at the time point of injection 2 and 3), 1 month after injection 3
  Quantitative parameter of red blood cells velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Kepler University Hospital, Linz, Austria